CLINICAL TRIAL: NCT03394105
Title: Pilot Study to Evaluate the Effect of Intrapleural Docetaxel Administration Using Medical Pleuroscopy in Malignant Effusion With Lung Cancer
Brief Title: Intrapleural Docetaxel Administration Using Medical Pleuroscopy in Malignant Effusion With Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Chang-Min Choi, associate professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2015-00353_Pleurodesis
Record Dates: First submitted 2017-10-09; First posted 2018-01-09 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Pleural Effusion, Malignant; Non-small Cell Carcinoma
Keywords: Pleurodesis
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intrapleural docetaxel administration (Experimental): Docetaxel will be administed to interpleural space using medical pleuroscopy in malignant effusion with lung cancer.
  Interventions: Drug: intrapleural docetaxel administration

INTERVENTIONS:
Drug: intrapleural docetaxel administration — intrapleural docetaxel administration using medical pleuroscopy in malignant effusion with lung cancer
  Other Names: Pleurodesis_docetaxel

SUMMARY:
In this trial, the effect of intrapleural docetaxel administration using medical pleuroscopywill be evaluated in Lung Cancer patient with malignant effusion.

DETAILED DESCRIPTION:
This study is designed to be pilot, single-center, open-label, single-arm, prospective, phase II trial of patient with NSCLC with pleurla effusion. Approximately 40 patients will be enrolled into the trial, and study will be performed to 31Dec2018 from IRB and Korea: MFDS approval date.

Docetaxel will be administed to interpleural space using medical pleuroscopy in malignant effusion with lung cancer. Response evaluation will be done until confiramtion of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20, and NSCLC patients with malignant pleural effusion and related symptoms
* ECOG ≤ 2
* Blood test ANC≥ 1500/mm3, Hb ≥ 8.0g/dl, platelet count ≥ 100000/mm3 Serum creatinine ≤ 1.8mg/dl, Total bilirubin within normal limits, Transaminases ≤ 1.5 x UNL, Alkaline phosphatase ≤ 2.5 X UNL BUN ≤ 25mg/dl, Creatinine clearance ≥ 50ml/min
* Negative serum or urine pregnancy test for women for childbearing age
* Patients who provide written informed consent for the study

Exclusion Criteria:

* Age < 20
* Patients who were previously perfomed pleurodesis
* Patients who were previously treated with thoracic radiosurgery
* Patinet with bilateral pleural effusion
* Age ≥ 80yrs
* Patients with histories of hypersensitivity to Docetaxel
* Patients with cardiovascular, respiratory, hepatic, renal, gastrointestinal, neunological disease, asthma, MI, stroke, arrhythmia, uncontrolled hypertionsion, etc. that would effect absorption, distribution, and metabolism of IP or be risk factors during IP administrion.
* Patients who could not understand the study procedure

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Overall respose rate(ORR) | through study completion (2.5 years)
  Rate of CR and PR
Complete resonse (CR) rate | through study completion (2.5 years)

SECONDARY OUTCOMES:
Time to progression(TTP) | through study completion (2.5 years)
  time from the date of the start of treatment until the disease progression or death.
Overall survival(OS) | through study completion (2.5 years)
  time fromthe date of the start of treatment to death or the date of last follow-up
Adverse Event | through study completion (2.5 years)
  Based on National Cancer Institute Common Toxicity Criteria

CONTACTS AND LOCATIONS:
Overall Officials: CHANG-MIN CHOI, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided